CLINICAL TRIAL: NCT00515346
Title: Phase 1 Study of Xpert(TM) Nitinol Stenting for Critically Ischemic Lower Limbs
Brief Title: Study to Evaluate the Safety & Performance of the Xpert(TM) Stent in Treating Below-the-knee Lesions in Patients Undergoing Percutaneous Intervention for Chronic CLI.
Acronym: XCELL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVA Physicians (Other)
Collaborators: Prairie Education and Research Cooperative (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060029
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Critical Limb Ischemia; Peripheral Vascular Diseases
Keywords: CLI; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Xpert(TM) Self-expanding Transhepatic Biliary Stent System feasibility in treating chronic critical limb ischemia

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the Xpert(TM) self-expanding stent in infrapopliteal lesions as part of an overall treatment strategy in patients undergoing percutaneous intervention for the treatment of documented chronic critical limb ischemia (CLI).

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) of the lower extremities affects roughly 25 million Americans annually. The diabetic population is particularly prone to the most severe clinical problems associated with PAD and the amputation rate amongst such patients is elevated five-fold. It has been shown that patients who undergo amputation for PAD/CLI have a much higher mortality rate in the months that follow.

Despite medical advances in the fields of pharmacology and wound care, the vast majority of patients who present with CLI will ultimately require amputation in the absence of improved blood flow. Recently, much attention has been directed towards less invasive endovascular solutions for treating patients with CLI. This study will evaluate approximately 140 subjects with Rutherford Class IV-VI PAD in a multi-center study in order to accurately estimate limb salvage rates for this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has documented wound care greater than or equal to 2 weeks prior to enrollment
* Subject understands the duration of the study and its follow up visit requirements
* Female subjects of childbearing potential have a negative pregnancy test less than 7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation
* Subject has documented chronic critical limb ischemia in the target limb for two weeks with Rutherford Category 4, 5 or 6
* Subject must have one of 5 approved non-invasive test results of the target limb within two weeks of enrollment.

Exclusion Criteria:

* Life expectancy of less than 12 months
* Cerebrovascular accident (CVA) or myocardial infarction (MI) within 3 months prior to enrollment
* Inability to walk (with assistance is accepted)
* Previous bypass surgery to target limb less than 30 days prior to study procedure
* Acute thrombus at the lesion site(s)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Amputation free survival at 12 months in the target limb. Amputation for the primary endpoint is defined as a major, unplanned, amputation of the target limb through the 12 month visit where prosthesis is required for standing or walking. | 1 year

SECONDARY OUTCOMES:
Assess improvement in wound healing; assess restenosis; measure target lesion revascularization to maintain patency at 12 months; measure ankle/brachial improvement level; assess stent integrity; characterize improvement in health related quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James D. Joye, DO, Principal Investigator — VIVA Physicians Inc.
Locations (1):
- VIVA Physicians Inc., San Jose, California, United States

REFERENCES:
- See also: Click here for more information about this study — http://www.prairieresearch.com/trial_XCELL_P.html